CLINICAL TRIAL: NCT03916835
Title: Pain Management Via Music Therapy During Cleaning Cares in Pediatric Intensive Care Unit
Brief Title: MUSIDORE PED Study
Acronym: MUSIDORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: UF 7654
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Pain Management; Music Therapy
Keywords: Pediatric Critical ill care or intensive care; anxiety; pain
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy during cleaning care 1 (Other): This group receives music therapy during cleaning care 1 and not during the cleaning care 2.
  Each patient will act as their own control
  Interventions: Device: Pain evaluation ( FLACC scale) before and during the cleaning care with and without music therapy.
- Music Therapy during cleaning care 2 (Other): This group receives music therapy during cleaning care 2 and not during the cleaning care 1.
  Each patient will act as their own control
  Interventions: Device: Pain evaluation ( FLACC scale) before and during the cleaning care with and without music therapy.

INTERVENTIONS:
Device: Pain evaluation ( FLACC scale) before and during the cleaning care with and without music therapy. — Each child will benefit two cleaning cares during hospitalization. One with music therapy and the other without music therapy.
  Every time, the preparation will be the same with an equipment installation in order to keep comparability and blind.
  Child will be videotaped without sound during the care. The order of music therapy intervention will be randomized.

SUMMARY:
The aim of this study is to measure the efficacy of music during a painful procedure in pediatric intensive care unit.

Music therapy has real effects on the pain level already proven in adults units. Our objective is to apply this technic to children. The investigators will evaluate this technic during cleaning care which is daily procedure for each stable patient and wich may be painful in this population.

DETAILED DESCRIPTION:
Pediatric intensive care units may be anxious places. A lot of painful and stressful procedures are done every day. A simple care such as a simple cleaning care may become painful or uncomfortable.

Usually those situation require the use of painkillers. For several years, new approaches are used in order to decrease the pain level without medication such as hypnosis or music therapy. Music therapy proved efficacy to reduce pain in different procedures and is currently used in adult intensive care units in order to decrease anxiety and pain.

One specific program, "Music Care" is based on a "U sequence" which use tempo and rhythm variations following the U scheme, to relax patients.

This program will be evaluated in our department and the investigators will study the effects on the pain level during a cleaning care .

The patients will be evaluated during two consecutive cleaning cares. One with and the other without music therapy. The investigators will compare the variation of the FLACC scores (before and during cleaning care ) to show a difference between both methods. The order (with or without) will be randomized. The patient will be his one control.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 6 months and 15 years old
* Vigil child
* Admitted to the department of Pediatric Critical Ill Unit at University Hospital in Montpellier (France)
* Signed both parental consent.
* Signed both parental authorization for videotape recording
* Parents or person with legal authority who speaks and understands french

Exclusion Criteria:

* Deaf child
* Refusal of the child to participate in the study

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
The FLACC (Face Legs Activity Cry Consolability) scale's score | Day 1 : 10 minutes before the care
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
The FLACC (Face Legs Activity Cry Consolability) scale's score | Day 1: During the care
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
The FLACC (Face Legs Activity Cry Consolability) scale's score | Day 2: 10 minutes before the care
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
The FLACC (Face Legs Activity Cry Consolability) scale's score | Day 2: During the care
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Cardiac frequency | Day 1 : 10 minutes before the care
  Values found on a device
Cardiac frequency | Day 1 : During the care
  Values found on a device
Cardiac frequency | Day 2 : 10 minutes before the care
  Values found on a device
Cardiac frequency | Day 2 : During the care
  Values found on a device
breathing frequency | Day 1: 10 minutes before the care
  Values found on a device
breathing frequency | Day 1: During the care
  Values found on a device
breathing frequency | Day 2: 10 minutes before the care
  Values found on a device
breathing frequency | Day 2: During the care
  Values found on a device
Mean arterial pressure | Day 1: 10 minutes before the care
  Values found on a device
Mean arterial pressure | Day 1: During the care
  Values found on a device
Mean arterial pressure | Day 2: 10 minutes before the care
  Values found on a device
Mean arterial pressure | Day 2: During the care
  Values found on a device
Duration care | Day 1
  Time management during cleaning cares
Duration care | Day 2
  Time management during cleaning cares

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Arnaud de Villeneuve- CHU Montpellier, Montpellier, France

REFERENCES:
- [Derived] Mounier S, Cambonie G, Baleine J, Le Roux M, Bringuier S, Milesi C. Music Therapy During Basic Daily Care in Critically Ill Children: A Randomized Crossover Clinical Trial. J Pediatr. 2024 Jan;264:113736. doi: 10.1016/j.jpeds.2023.113736. Epub 2023 Sep 16. PMID 37722559